CLINICAL TRIAL: NCT01647360
Title: A Post- Marketing, Prospective,Multicenter, Observational Program: Severity of Bleeding as a Predictor of Quality of Life (QoL) in Women With Heavy Menstrual Bleeding (HMB) Under Dydrogesterone Treatment
Brief Title: Severity of Bleeding as a Predictor of Quality of Life (QoL) in Women With Heavy Menstrual Bleeding (HMB) Under Dydrogesterone Treatment
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: P13-699
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Menorrhagia; Metrorrhagia
Keywords: Metrorrhagia; Menorrhagia
MeSH Terms: conditions — Menorrhagia; Metrorrhagia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women with Heavy Menstrual Bleeding (HMB)

SUMMARY:
Dydrogesterone is a retroprogesterone with a molecular structure similar to natural progesterone. As a C-21 steroid, it has a high affinity for progesterone receptors, a low antigonadotropic activity and antiestrogenic activity, but almost no estrogenic or androgenic activity. Dydrogesterone (Duphaston©) is indicated for dysfunctional bleeding.

In this study, women suffering from menorrhagia and who are treated with dydrogesterone will be observed for impact on QoL with the reduction in severity of bleeding.

ELIGIBILITY:
Inclusion Criteria

* Females aged 18 to 45 years
* Subjects presenting with Heavy Menstrual Bleeding (HMB)
* Subjects with Pictorial Blood Assessment Chart (PBAC) score of 100 or more
* Subjects will be treated with dydrogesterone in accordance to the local label after enrollment in the trial

Exclusion Criteria

* Subjects with structural or organic pathology as an underlying cause of HMB.
* Subjects with hypersensitivity to dydrogesterone
* Known or suspected progestogen dependent neoplasms
* Subjects with vaginal bleeding who have not been screened for organic or structural pathology as an underlying cause
* Subjects with acute or chronic liver disease
* Patients with depressive illness
* Subjects who are known to have rare hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* Nursing mothers
* Use of any other medication for uterine bleeding (including but not limited to progesterone, oral contraceptive pills, tranexamic acid etc)
* Use of Non-Steroidal Anti inflammatory Drugs (NSAIDs)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with heavy menstrual bleeding
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
EQ-5D Quality of Life questionnaire | 3 months
  The EQ-5D assesses five dimensions of HRQOL: mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each dimension is measured on a three-point ordinal scale where a higher score corresponds to a worse health state (no limitation, some limitation, and greatest limitation in HRQOL). This will be evaluated at baseline and then at each follow up visit to see impact on quality of life.

SECONDARY OUTCOMES:
Pictorial Blood Assessment Chart (PBAC) score | 3 months
  PBAC score of 100 or more corresponds with heavy menstrual bleeding. PBAC score will be assessed at each visit to see any improvement.
Menstrual Cycle Diary | 3 months
  Change in the nature of menstruation will be taken into account based on the subjects' perception as recorded on the Menstrual Cycle Diary.

CONTACTS AND LOCATIONS:
Overall Officials: Raeef Ahmed, MD, Study Director — Abbott
Locations (20):
- Pakistan (20):
  - Site reference ID/Investigator# 79836, Islamabad, Federal Capital
  - Site Reference ID/Investigator# 77674, Karachi, Sindh
  - Site Reference ID/Investigator# 77675, Karachi, Sindh
  - Site reference ID/Investigator# 77676, Karachi, Sindh
  - Site Reference ID/Investigator# 77677, Karachi, Sindh
  - Site Reference ID/Investigator# 77680, Karachi, Sindh
  - Site Reference ID/Investigator# 77681, Karachi, Sindh
  - Site reference ID/Investigator # 77690, Lahore, Punjab
  - Site Reference ID/Investigator# 77691, Lahore, Punjab
  - Site reference ID/Investigator# 77694, Lahore, Punjab
  - Site Reference ID/Investigator# 77695, Lahore, Punjab
  - Site Reference ID/Investigator# 77696, Lahore, Punjab
  - Site reference ID/Investigator# 77698, Lahore, Punjab
  - Site Reference ID/Investigator# 77699, Lahore, Punjab
  - Site Reference ID/Investigator# 77686, Multan, Punjab
  - Site Reference ID/Investigator# 77687, Multan, Punjab
  - Site Reference ID/Investigator# 77684, Multan, Punjab
  - Site Reference ID/Investigator# 77689, Multan, Punjab
  - Site reference ID/Investigator # 77693, Rawalpindi, Punjab
  - Site reference ID/Investigator# 79834, Rawalpindi, Punjab